CLINICAL TRIAL: NCT03386565
Title: Effect of Intraoperative IV Lidocaine Infusion on Intraoperative Isoflurane Requirements
Brief Title: Effect of Intraoperative Lidocaine Infusion on Intraoperative Isoflurane Requirements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed galal aly, Assistant Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1720147
Record Dates: First submitted 2017-12-17; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sodium Chloride; Saline Solution; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): * Sodium chloride solution 10 mL IV just before induction of anesthesia
  * IV infusion during the surgery
  Interventions: Drug: sodium chloride solution
- lidocaine group (Active Comparator): * lidocaine 2 mg ̸ kg slowly IV just before induction of anesthesia
  * IV infusion during the surgery
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: sodium chloride solution — intraoperative IV infusion
  Other Names: normal saline solution
  Arms: control group
Drug: Lidocaine — intraoperative IV infusion
  Other Names: xylocaine
  Arms: lidocaine group

SUMMARY:
Fifty patients were included in the study, divided into two equal groups (25 in each), underwent spinal fusion surgery.Control group: received normal saline.

Lidocaine group: received lidocaine 2.0 mg/kg slowly IV before induction of anesthesia, followed by lidocaine IV infusion at a rate of 2.5 mg/kg/hr until the end of surgery. We evaluated the end-tidal isoflurane concentration required to maintain AAI index in the range of 20-25 during adult spinal fusion surgery.

DETAILED DESCRIPTION:
This prospective, double-blinded, randomized study was carried out in Assiut University Hospitals, after approval by the local research ethics committee of Assiut Faculty of Medicine, Egypt. Informed consent was taken from each patient.

Patients were randomly allocated into two groups of equal size to receive either 0.9% sodium chloride infusion group 1 (CG), or lidocaine infusion group 2 (LG). Randomization was performed using G1 and G2 registers, which was placed in sealed envelopes prior to study initiation and opened prior to anesthesia by a physician who prepared the intravenous solution and identified it with the patient number, according to the envelope drawn. The solution was handed to another physician, blind to the prepared solutions' content, who was responsible for the anesthesia. The solution volume was equal. The responsible investigator was remained blind to the chosen group until the end of the study. G1 patients (n = 25) were received 10 mL of 0.9% sodium chloride slowly IV just before induction of anesthesia, then infused through 50 mL syringe as lidocaine, and G2 patients (n = 25) were received a loading dose of lidocaine 2 mg ̸ kg (maximally 200 mg) slowly IV just before induction of anesthesia, then the lidocaine infusion started immediately after positioning at a rate of 2.5 mg ̸ kg/h until the end of the procedure (50 mL syringe contained 25 mL 2.0% lidocaine i.e., 500 mg lidocaine plus 25 mL normal saline). Both syringes (10 mL for loading dose and 50 mL for maintenance IV infusion) were labelled by the case number and prepared by another anesthesiologist who did not share in anesthesia.

Anesthesia technique: Patients were monitored with continuous electrocardiography, pulse oximetry and intermittent non-invasive blood pressure measurements every 5 min. Capnography, end-tidal isoflurane concentration (Et-Iso) via AVANCE CS2 Datex-Ohmeda, Inc. USA, and auditory evoked potential monitor (AEP monitor 2 Dia Trade medical engineering) also attached to the patient (one AEP electrode was placed on the center of the forehead, one on the temple, and one behind the left ear over the mastoid bone).

General anesthesia was induced by propofol 2.5 mg ̸ kg and cisatracurium 0.15 mg ̸ kg to facilitate endotracheal intubation. Patients were then assigned to two groups by closed-envelope randomization. In both groups, anesthesia was maintained with isoflurane in oxygen/air mixture at sufficient concentration to maintain AAI index in the range 20-25, and mean blood pressure within 25% of the baseline value. All patients were received 60 mg ketorolac (ketolac) slowly IV after induction of anesthesia, and fentanyl 1.5 µg ̸ kg IV before skin incision and 0.5 µg ̸ kg given IV after 45 min. Reversal of residual muscle relaxant was done using neostigmine and atropine at the end of the operation.

Data collection: Demographic and surgical data include: Age, gender, weight, height, duration and type of surgery, in addition to Et-Iso.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients underwent spinal fusion surgery ASA I, II and III

Exclusion Criteria:

* History of epilepsy hearing disorders known allergy to lidocaine BMI > 35 significant cardiac diseases significant renal diseases liver dysfunction substance abuse chronic opioid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10-02 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
effect of intraoperative IV lidocaine infusion on intraoperative end tidal isoflurane concentration | every 15 minutes from induction of anesthesia until 90 minutes intraoperative.
  using gas analyzer for determination of end tidal isoflurane concentration (%) (ET-Iso) needed to maintain AAI index in the range 20-25.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vesal N, Spadavecchia C, Steiner A, Kirscher F, Levionnois OL. Evaluation of the isoflurane-sparing effects of lidocaine infusion during umbilical surgery in calves. Vet Anaesth Analg. 2011 Sep;38(5):451-60. doi: 10.1111/j.1467-2995.2011.00636.x. PMID 21831050
- [Background] Saadawy IM, Kaki AM, Abd El Latif AA, Abd-Elmaksoud AM, Tolba OM. Lidocaine vs. magnesium: effect on analgesia after a laparoscopic cholecystectomy. Acta Anaesthesiol Scand. 2010 May;54(5):549-56. doi: 10.1111/j.1399-6576.2009.02165.x. Epub 2009 Nov 16. PMID 19919581